CLINICAL TRIAL: NCT01712711
Title: The Effect of Helicobacter Pylori Eradication on Liver Fat Content in Diabetic Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: Helicobacter Pylori Eradication in Diabetic Subjects With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Raika Jamali, MD, Assistant Professor of Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1391/7/24-579
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Steatohepatitis,; Helicobacter pylori,; Insulin resistance,; Alanine aminotransferase,; Aspartate aminotransferase,
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Insulin Resistance

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle modification (No Intervention): Obtaining ideal body weight by calorie restriction diet and programmed physical activity
- H.pylori eradication (Experimental): H.pylori eradication by quadruple antibiotic therapy for two weeks plus obtaining ideal body weight by calorie restriction diet and programmed physical activity
  Interventions: Drug: H.pylori eradication

INTERVENTIONS:
Drug: H.pylori eradication — The regimen consists of Omeprazole (20 mg/BD)+ Amoxicillin (1 g/day)+ Bismuth subcitrate (240 mg/BD)+ Azithromycin (500 mg/BD)for two weeks
  Other Names: Helicobacter pylori treatment
  Arms: H.pylori eradication

SUMMARY:
The aim of study was to evaluate the effect of helicobacter pylori eradication on liver fat content, liver function tests, lipid profile, homeostasis model assessment-IR (HOMA-IR) index, and anthropometric measurements (body mass index and waist circumference)in diabetic subjects with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Helicobacter pylori (HP) antigens have been found in the liver of individuals with benign and malignant liver diseases. The role of HP in the pathogenesis of non-alcoholic fatty liver disease (NAFLD) is controversial.

This randomized double blind clinical trial was performed in diabetic dyspeptic patients with positive antibody to HP and the evidence of fatty liver in ultrasonography. After excluding other causes, participants with persistent elevated serum aminotransferase levels were presumed to have NAFLD. Those with NAFLD liver fat score greater than (-0.64) and positive urea breath test (UBT) were enrolled. They were randomly assigned to lifestyle modification alone or lifestyle modification plus HP eradication groups. Quadruple therapy (omeprazole, amoxicillin, bismuth subcitrate, and clarithromycin) for HP eradication was performed in two weeks. HP eradication was documented by UBT. Liver fat content, fasting serum glucose, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, triglyceride, cholesterol, high and low-density lipoprotein, HOMA-IR, and anthropometric measurements (body mass index and waist circumference) were checked at baseline and six weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic dyspeptic patients with positive antibody to H.pylori and persistent elevated aminotransferase levels with the evidence of fatty liver in ultrasonography, who were referred to a gastroenterology clinic

Exclusion Criteria:

* Alcohol use (more than 20 gram per day in men and 10 gram per day in women per day), heart disease (ischemic or congestive), hepatic disease (viral hepatitis, autoimmune hepatitis, wilson disease, hemochromatosis, liver mass lesion), renal disease (serum creatinine concentration of > 1.5 mg/dl), any severe systemic co-morbidities, neoplasm, using any hepatotoxic medication during the past 3 months, previous history of peptic ulcer, previous history of H.pylori eradication, existence of alarm signs (weight loss, dysphagia, anemia, vomiting, positive family history of gastrointestinal cancers), and pregnant or lactating women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raika Jamali, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Gastroenterology clinic, Sina Hospital, Tehran, Iran

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Modification | H.Pylori Eradication
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Modification | H.Pylori Eradication | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.95 (9.53) | 45.73 (12.54) | 42.84 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 12 | 8 | 20
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Liver Fat Content Change From Baseline to Six Weeks Post H.Pylori Treatment
Description: Liver fat content was calculated by a valid formula. The formula is as the followings:Liver fat content (%) = 10 (-0.805 + 0.282 * metabolic syndrome (yes = 11 no = 0) + 0.078 * type 2 diabetes (yes =2 / no =0) + 0.525 * log fasting serum insulin (mU/L) + 0.521 * log fasting serum AST (U/L) - 0.454 * log (AST/ALT)
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of liver fat content
Arm/Group | Lifestyle Modification | H.Pylori Eradication
Number analyzed (Participants) | 20 | 20
percentage of liver fat content | 2.46 (2.23) | 3.61 (3.25)

ADVERSE EVENTS:
Time Frame: 1 year
Description: self-reporting by participants
Arm/Group | Lifestyle Modification | H.Pylori Eradication
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
No limitation existed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes